CLINICAL TRIAL: NCT01786655
Title: Neosaxitoxin (NeoSTX) Alone and in Combination With Bupivacaine as Prolonged Duration Local Anesthetics: A Phase I Investigator-initiated Dose Escalation Study
Brief Title: Safety Study of Long-Acting Local Anesthetic
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Charles Berde (Other)
Responsible Party: Sponsor-Investigator, Charles Berde, Chief, Division of Pain Medicine (Department of Anesthesiology, Perioperative, and Pain Medicine), Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: IRB-P00003344
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Safety of Neosaxitoxin in Healthy Volunteers
Keywords: local anesthetic; neosaxitoxin; neoSTX; bupivacaine; safety; phase 1; pharmacokinetic
MeSH Terms: interventions — neosaxitoxin; Sodium Chloride; Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Neosaxitoxin in saline (Experimental): Subjects receive only one injection of NeoSTX in saline on the back of one calf (test side). Subjects receive NeoSTX in saline in subsequent dose escalation levels: 5mcg, 10mcg, 15mcg, 20mcg, 30mcg, and 40mcg NeoSTX.
  Interventions: Drug: Neosaxitoxin in saline
- Neosaxitoxin + bupivacaine 0.2% (Experimental): Subjects receive only one injection of NeoSTX in combination with 0.2% bupivacaine on the back of one calf (test side). Subjects receive NeoSTX in bupivacaine in subsequent dose escalation levels: 5 mcg, 10 mcg, 15 mcg, 20 mcg, 30 mcg, and 40 mcg NeoSTX.
  Interventions: Drug: NeoSTX + bupivacaine 0.2%
- Neosaxitoxin + bupivacaine 0.2% + epinephrine 5mcg/ml (Experimental): Subjects receive one injection of NeoSTX in bupivacaine 0.2% with epinephrine 5 mcg/ml on the back of one calf (test side). Subjects receive NeoSTX in bupivacaine 0.2% with epinephrine 5 mcg/ml in doses of 10 mcg or 30 mcg of NeoSTX.
  Interventions: Drug: NeoSTX + bupivacaine 0.2% + epinephrine 5mcg/ml
- Saline placebo (Placebo Comparator): Subjects receive one injection of saline on the back of one calf (test side).
  Interventions: Other: Saline placebo

INTERVENTIONS:
Drug: Neosaxitoxin in saline — NeoSTX will be administered in sequential dose cohorts. Each subject receives one injection with bupivacaine 0.2% alone on one side (control). On the other side they receive NeoSTX in saline (test). Subjects receive NeoSTX in saline in subsequent dose escalation levels: 5 mcg, 10 mcg, 15 mcg, 20 mcg, 30 mcg, and 40 mcg of NeoSTX.
  Arms: Neosaxitoxin in saline
Drug: NeoSTX + bupivacaine 0.2% — NeoSTX will be administered in sequential dose cohorts. Each subject receives one injection with bupivacaine 0.2% on one side (control). On the other side they receive NeoSTX with 0.2% bupivacaine. Subjects receive NeoSTX in 0.2% bupivacaine in subsequent dose escalation levels: 5 mcg, 10 mcg, 15 mcg, 20 mcg, 30 mcg, and 40 mcg of NeoSTX.
  Arms: Neosaxitoxin + bupivacaine 0.2%
Drug: NeoSTX + bupivacaine 0.2% + epinephrine 5mcg/ml — Each subject receives one injection with bupivacaine 0.2% on one side (control). On the other side they receive NeoSTX in 0.2% bupivacaine with epinephrine 5 mcg/ml. Subjects receive NeoSTX in 0.2% bupivacaine with epinephrine 5 mcg/ml in doses of 10 mcg or 30 mcg of NeoSTX.
  Arms: Neosaxitoxin + bupivacaine 0.2% + epinephrine 5mcg/ml
Other: Saline placebo — Each subject receives one injection with bupivacaine 0.2% alone on one side. On the other side they receive saline placebo.
  Arms: Saline placebo

SUMMARY:
The primary aim of this Phase 1 study is to evaluate the systemic safety of a novel prolonged-duration local anesthetic, Neosaxitoxin (NeoSTX), given by subcutaneous injection in combination with the commonly used local anesthetic, bupivacaine, and epinephrine.

The investigators hypothesize that a "minimal adverse effect threshold" NeoSTX dose for subcutaneous administration in combination with bupivacaine 0.2% and epinephrine 5mcg/ml respectively, can be defined for awake, young adult healthy volunteer subjects. At the same time, the pharmacokinetics of NeoSTX when delivered subcutaneously will be determined.

DETAILED DESCRIPTION:
Currently available amino amide local anesthetics (e.g. bupivacaine, levobupivacaine, ropivacaine) do not reliably provide analgesia beyond roughly 8 hours following subcutaneous infiltration. In addition, they can cause systemic toxicities such as seizures, arrhythmias, and cardiac arrest, as well as local tissue toxicities to muscle, cartilage and nerve. Therefore, there is a need for safe local anesthetics that can provide longer duration analgesia with low systemic and local tissue toxicities.

The investigator team previously reported that tetrodotoxin, saxitoxin, and NeoSTX could produce prolonged sensory blockade (numbness) and motor blockade (weakness) following injection near the sciatic nerves in rats. In these studies, combining the site 1 toxin with either bupivacaine or epinephrine dramatically improved efficacy (duration of sensory blockade) and reduced systemic toxicity.

NeoSTX is the most potent member of the STX series identified to date. In preliminary studies, investigators at the University of Chile, Santiago, and with a small biotech company, Proteus S.A, developed a bioreactor process to produce clinical grade NeoSTX efficiently, with excellent purity, stability, sterility and non-pyrogenicity. A series of preclinical safety and toxicologic studies in mice, rats, and sheep were performed at CHB and Toxikon, Inc.

In this proposal, the investigators plan to conduct a Phase I study to be performed under an Investigator-Initiated FDA IND to further establish the systemic and local safety of escalating doses of NeoSTX via sub-cutaneous infiltration in healthy and awake young adult male human volunteer subjects.

The primary aim of this Phase 1 study is to evaluate the systemic safety of a novel prolonged-duration local anesthetic, neosaxitoxin (NeoSTX), given by subcutaneous injection, either alone or in combination with the commonly used local anesthetic, bupivacaine, and epinephrine. The hypothesis is that, using adverse events as endpoints, a "minimal adverse effect threshold" NeoSTX dose for subcutaneous administration in combination with bupivacaine 0.2% and epinephrine 5mcg/ml respectively, can be defined for awake, young adult healthy volunteer subjects.

In double blind fashion, each subject will receive two injections simultaneously in a 3 cm x 3cm square area on skin of the posterior aspect of the lower leg (calf), one on each side. Each subject receives one injection with bupivacaine 0.2% alone on one side. On other side, they will receive one of 4 possible solutions: (1) saline placebo, (2) NeoSTX in saline or (3) NeoSTX in combination with bupivacaine or (4) NeoSTX in combination with bupivacaine 0.2% and epinephrine 5mcg/ml.

In each dose group, only one of the injections involves placebo. Prior to each dose increase, there is a safety review and confirmation that no stopping rule has been reached.

Specific Aims

1. Measure the dose dependence of FDA-AEs and SD-AEs from NeoSTX in saline;
2. Measure the dose dependence of FDA-AEs and SD-AEs from NeoSTX in bupivacaine 0.2%;
3. Measure the dose dependence of FDA-AEs and SD-AEs from NeoSTX in bupivacaine 0.2% with epinephrine 5mcg/ml;
4. Measure the serum and urine concentrations of NeoSTX following injections of NeoSTX alone or with bupivacaine 0.2% with and without epinephrine; and correlate the serum concentrations with the "Systemic Effects";
5. Evaluate skin integrity and other potential local reactions (edema, numbness, and paresthesia, erythema) in treated limbs receiving NeoSTX-saline, NeoSTX-bupivacaine, NeoSTX-bupivacaine-epinephrine or plain bupivacaine.
6. Using QST, establish the dependence of sensory blockade intensity and duration on NeoSTX dose and on presence or absence of bupivacaine and epinephrine;

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males ages 18-35
2. ASA physical status 1 or 2
3. English or Spanish speakers
4. Must be able to come to Boston Children's Hospital for a 24-hour stay and able and willing to attend 5-10 study visits
5. Must be able to provide informed consent
6. Must be able to understand and perform all the procedures of the study including self-reporting of symptom scores

Exclusion Criteria:

1. ASA physical status 3 or greater
2. Cognitively challenged or other inability to understand the self-report measures or to give informed consent
3. Significant cardiovascular, respiratory, neuromuscular disease or other systemic illness(es)
4. No known or suspected allergies to neosaxitoxin, bupivacaine, or other local anesthetics
5. Subjects may not be on any pain controlling medications, or any medications that would alter pain tolerance
6. Subjects may not be on any medication that would alter cognition
7. Subjects may not have any acute or chronic pain conditions requiring ongoing treatment or limiting daily activities
8. No alcohol or illicit drug abuse
9. No current smokers

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Presence or absence of Adverse Events as a function of NeoSTX dose | Within 14 days of injection

SECONDARY OUTCOMES:
Pharmacokinetic parameters characterizing uptake and distribution of NeoSTX (content in serum and urine samples) | Within 24 hours of injection
Cutaneous sensory blockade (numbness) | Within 14 days of injection
  measured by noninvasive quantitative sensory testing (QST)
Local skin reactions (edema, paresthesias and urticaria) | Within 14 days of injection

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cravero, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States